CLINICAL TRIAL: NCT04412746
Title: Prevalence of Diabetes Among Hospitalized Patients With Covid-19 in West of Algeria. Identification of Diabetes-related Associated Factors Severe Forms
Brief Title: Covid-19 and Diabetes in West of Algeria
Acronym: COVIDIAB-13
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laboratoire De Recherche Sur Le Diabete, Université de Tlemcen (Network)
Collaborators: ATRSS, DGRST, Algeria (Unknown)
Responsible Party: Principal Investigator, ALI LOUNICI, Chief of Internal Medicine Department, Laboratoire De Recherche Sur Le Diabete, Université de Tlemcen
Other Study IDs: COVIDIAB-13
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infections; Diabetes Mellitus; Prevalence; Risk Factors; Patient Outcome Assessment; Severe Acute Respiratory Syndrome
Keywords: COVID-19; DIABETES; RISK FACTORS; SEVERE ILLNESS; OUTCOMES
MeSH Terms: conditions — Coronavirus Infections; Diabetes Mellitus; Severe Acute Respiratory Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: MANAGEMENT OF COVID-19 — MANAGEMENT OF COVID-19 Oxygen therapy to maintain SpO2 target more than 94%. Low molecular weight heparin (LMWH) at preventive doses. Empirical antibiotic treatment.
  Specific treatment for COVID-19 (approved by Algerian Ministry of Health) First line: Hydroxychloroquin: 200 mg oral three times a day for 10 days, with association of Azithromycin 250 mg oral : 500 mg the first day and 250 mg once a day for 4 days. Sulfate de Zinc : 220 mg once a day for 5 days. Second line: Lopinavir/ritonavir capsule 200 mg/50 mg, oral 2 capsules each times, twice a day during 5 to 7 days.
  IF AGGRAVATION OR CRITICAL ILL CONDITION AT PRESENTATION Increase oxygenation flow. Consider Glucocorticoids. 3. Consider the diagnosis of pulmonary embolism and treat with LMWH at therapeutic doses.
  MANAGEMENT OF DIABETES Discontinue metformin. Start or adjust insulin doses according to personalized glycemic target of patient.
  Other Names: MANAGEMENT OF DIABETES

SUMMARY:
By Jan 7, 2020, Chinese scientists had isolated a novel coronavirus, from patients with virus-infected pneumonia. The WHO designated later this virus as COVID-19 (coronavirus disease 2019). This exponential pandemic coronavirus infection is responsible for severe forms in 15 to 20%, for critical ill requiring ventilation in 5% and for mortality in 2%. Algeria was part of the 13 top priority countries identified by WHO based on their direct links and volume of travel to the infected provinces in China.

It is known that some predisposing conditions lead to a worse outcome with coronavirus.

In China, the overall case-fatality rate was 2.3%, but was higher in patients with diabetes (7.3%). In Italy, the most common comorbidities associated with death from COVID-19 were hypertension (73.8%) and diabetes (33.9%). The US Centers for Disease Control and Prevention suggests diabetes is the most common comorbidity in COVID-19 cases. In the largest cohort NHS England study, death from COVID-19 was strongly associated with uncontrolled diabetes (after full adjustment, HR 2.36).

The West Algerian CORODIAB-13 study aims is (1) to assess the prevalence of diabetes among hospitalized patients with Covid-19, (2) to describe the phenotypic characteristics of patients with diabetes, and (3) to identify the parameters specific to the diabetic which are associated with severe forms.

In the future, this study will provide answers for two main questions

1. Why diabetics are more at risk of developing Covid-19 infection?
2. Why diabetics are at high risk of developing severe forms?

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in a hospital center since 1th April 2020
* Patients with COVID19 with biological proof (specific PCR) or with clinical and radiological diagnosis.
* Patient with diabetes known before the admission
* New onset diabetes discovered at admission (plasma glycaemia value strictly greater than 2 g/l at any time)

Exclusion Criteria:

* Pregnant
* Active Cancer
* Dementia
* Minors, adults under guardianship, protected persons
* Significant disability (The Modified Rankin Scale more than 2 prior admission)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults diabetic patients with COVID-19 infection admitted in academic hospital of Tlemcen (Algeria).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diabetes among all hospitalized COVID-19 | 3 months
  Assess the prevalence of diabetes among hospitalized patients with Covid-19 in Area of Tlemcen
Diabetes-related factors risk | 3 months
  Describe the clinical and biological characteristics of hospitalized subjects with diabetes and COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Acedemic Hospital of Tlemcen, Tlemcen, Algeria

IPD SHARING:
Plan to Share IPD: No